CLINICAL TRIAL: NCT07334704
Title: Effects of Implementing a Program to Develop Emotional Skills and Post-traumatic Growth in Adolescents and Young Adults Receiving Child Welfare Services-a Pilot Study in the Haute-Loire Department
Acronym: JEMotion43
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Emile Roux (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: RIPH3_PEREIRA_JEMotion43
Record Dates: First submitted 2025-12-31; First posted 2026-01-12 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Child Protection Service; Child Welfare
MeSH Terms: interventions — Surveys and Questionnaires; Restraint, Physical

STUDY DESIGN:
Intervention Model Description: Pilot study, RIPH 3, controlled and non-randomized, with two parallel arms and a mixed methodological approach (quantitative and qualitative).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Participation in a structured 6-week program focused on emotional skills development and psychoeducation on post-traumatic growth (JEMotion43 program).
  Interventions: Other: Questionnaire and Physical Exam; Other: Program JEMotion
- Control Group (Active Comparator): Use, over the same period, of a mobile app promoting mental health (WeCare / Care Island).
  Interventions: Other: Questionnaire and Physical Exam; Other: mobile app

INTERVENTIONS:
Other: Questionnaire and Physical Exam — completion of all questionnaires :
  * l'Adverse Childhood Experiences-International Questionnaire
  * Benevolent Childhood Experiences
  * Emotional Competency Profile
  * psychological distress (K6)
  * Warwick-Edinburgh Mental Well-Being Scale
  * Post traumatic Growth Inventory
  * Attention Assessment Tests
  * Wechsler Adult Intelligence Scale
  * Behavior Rating Inventory of Executive Function
Other: Program JEMotion — Programm JEMotion : 6-week emotional skills development and psychoeducation program. It consists of 8 modules of 2 hours each.
  The program is structured around a variety of activities based on pedagogical and experiential principles. It includes enriching emotional vocabulary, identifying emotional components, and exploring their functional value.
  Arms: Intervention Group
Other: mobile app — Mobile app promoting mental health for teens aged 14 to 17. It is a gamified, self-guided 6-week digital program (about 1 hour per week), incorporating techniques from cognitive behavioral therapy, positive psychology, and lifestyle medicine.
  The game offers a narrative journey through an imaginary world consisting of six islands, each corresponding to a health and well-being theme: physical activity, stress management, sleep, addictive behaviors, emotional regulation, automatic thoughts, and self-compassion. Side quests also address balanced eating and the integration of positive psychology practices into everyday life.
  The player takes on the role of a hero accompanied by their guide, tasked with restoring the vital balance of the islands threatened by pollution and destruction. The player must clean up the islands, recycle waste into seeds, regenerate nature, and interact with totem animals, which impart psychoeducational lessons related to mental health.
  Arms: Control Group

SUMMARY:
Adolescents and young adults receiving child welfare services constitute a vulnerable population, with an overrepresentation of mental health issues and past trauma, often exacerbated by a difficult transition to independence. Current support focuses mainly on material needs, lacking specific interventions targeting psychological resilience. This study draws on literature demonstrating that the development of emotional skills and post-traumatic growth are major protective factors promoting psychosocial adaptation and mental health.

ELIGIBILITY:
Inclusion Criteria:

* Minors: > 15 to < 18 years old:

  1. Be taken in or accompanied by a child protection service.
  2. Have given informed consent to participate in the study.
  3. Have obtained authorization from those with parental authority.

Young adults aged ≥ 18 to 21:

1. Have signed a young adult contract (CJM) with the Child Welfare Service (ASE).
2. Have given their informed consent to participate in the study.

Ages: 15 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 32 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-09 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Emotional Competence | Baseline and 6 months
  score assessed by Emotional Skills Profile. 45 items from this instrument assess the management of one's own emotions. 15 subscale covers five skills : identifying, understanding, expressing, regulating, and using emotions, over 3 targets : self / others / context Each item is rated on a 5-point Likert scale. The total ESP score ranges from 45 to 225 (45 items rated from 1 to 5) and reflects the overall level of emotional skills, with a low score indicating poorly developed skills, a medium score indicating adequate emotional functioning, and a high score indicating good abilities to identify, express, regulate, and use emotions.
post-traumatic growth | Baseline and 6 months
  Score assessed by Posttraumatic Growth Inventory (PTGI) This 21-item questionnaire measures perceived positive psychological changes following adversity. It covers five dimensions: relationships with others, personal strength, new possibilities, spiritual changes, and appreciation of life.
  The score is calculated by adding up the scores for the 21 items (rated from 0 = no change to 5 = very significant change), giving a total score between 0 and 105. Subscale scores can also be obtained by adding up the items corresponding to each of the five dimensions.
  A low score indicates little perceived positive change after the event, a moderate score indicates partial growth, and a high score indicates significant positive psychological transformation.

SECONDARY OUTCOMES:
Mental well-being | Baseline, 1 week before intervention and 6 months
  Mental well-being will be assessed using the Warwick-Edinburgh Mental Well-Being Scale.The total WEMWBS score ranges from 14 to 70 and reflects the overall level of mental well-being, with a low score indicating reduced well-being, a medium score indicating moderate well-being, and a high score indicating significant and positive mental well-being.
Psychological distress | Baseline, 1 week before intervention and 6 months
  Psychological distress will be measured using the French version of the Kessler Brief Symptom Inventory (K6). This 6-item self-report questionnaire assesses the frequency of nonspecific emotional distress symptoms (e.g., feeling "nervous" or "despairing") over the past 30 days. Responses are given on a 5-point scale indicating frequency (from "Never" to "All the time"). To calculate the score, responses are rated from 0 to 4, generating a total score ranging from 0 to 24, where a higher score indicates greater distress.
executive functions | Baseline, 1 week before intervention and 6 months
  The Behavioral Rating Inventory of Executive Functions is a self-assessment questionnaire for executive functions. It comprises 75 items assessing 9 areas of executive functions. The total score is expressed as a T-score (mean 50, standard deviation 10) and reflects the overall level of executive functioning, with a T-score ≥ 65 indicating significant difficulties, T 60-64 indicating a borderline area, and T < 60 indicating average executive functioning.
Attention | Baseline, 1 week before intervention and 6 months
  The Attention Assessment Tests score is summarized by standardized scores or percentiles for each domain (sustained, divided, selective attention, and motor inhibition), reflecting overall attentional performance, where high scores indicate adequate attention and executive control, and low scores reveal specific difficulties in one or more aspects of attention.
working memory | Baseline, 1 week before intervention and 6 months
  The ARITHMETIC and NUMBER MEMORY subtests of the Wechsler Adult Intelligence Scale can be used to assess working memory. The Working Memory Index, based on the Arithmetic and Number Memory subtests, is expressed as a standard score (mean 100, standard deviation 15 for the overall index, or 10/3 for the subtests) and reflects working memory capacity, where a low score indicates difficulties in maintaining and manipulating information, an average score indicates expected functioning, and a high score indicates above-average working memory.

CONTACTS AND LOCATIONS:
Overall Officials: Mathieu PEREIRA, Principal Investigator — Université Lumière Lyon 2